CLINICAL TRIAL: NCT05876988
Title: The Role of Chinese Acupuncture for Chemotherapy Induced Cognitive Impairment in Elderly Cancer Patients
Brief Title: Chinese Acupuncture for Chemobrain in Elderly Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Jiangsu Health Vocational College (Unknown)
Responsible Party: Principal Investigator, Gong yongling,MD, PI, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nanjing First
Record Dates: First submitted 2023-04-13; First posted 2023-05-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Chinese Acupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Electroacupuncture intervention will take about 45 minutes every time. For experimental group, acupuncture points are mainly in the head, limbs and abdomen, and a total of six pairs of electric acupuncture for head. The Montreal Cognitive Assessment (MoCA) serves as the primary outcome. Digit span test will be the secondary outcome for attentional function and working memory. In addition, EORTCQLQ-C30 will be used to examine the quality of life of elderly cancer patients. Functional changes and side eﬀects associated with therapies will be measured using the Functional Assessment of Cancer Therapy (FACT). Most items of these functional assessments are 5-point Likert scale questions. Functional items which would be rated as "3" (quite a bit) or higher and incidences would be signiﬁcantly diﬀerent between the two groups in any assessment point will be extracted for statistical analysis.
  Interventions: Device: Chinese acupuncture
- control group (Placebo Comparator): Electroacupuncture intervention will take about 45 minutes every time. For the control group, acupuncture points are mainly on the head and limbs, only a pair of electric needles for head. The Montreal Cognitive Assessment (MoCA) serves as the primary outcome. Digit span test will be the secondary outcome for attentional function and working memory. The quality of life and multiple functional assessments will also be evaluated.
  Interventions: Device: Chinese acupuncture

INTERVENTIONS:
Device: Chinese acupuncture — Disposable acupuncture needles(0.30mm in diameter and 25-40mm in length) will be inserted at a depth of 10-30mm perpendicularly or obliquely into acupoints. Manual manipulation will be carried out for all acupoints to evoke needling sensation. Electrical stimulation was additionally delivered on the 6 pairs of the frontal acupoints. The output peak current and voltage of the machine would be 6V and 48mA, respectively, with constant wave at frequency of 2Hz and phase duration of 100µs for 30min. Electrical stimulation lasted 30min. The needles on body acupoints will be also retained for 30min.
  Acupuncture intervention will be conducted for 2 sessions per week over 8 consecutive weeks. The determination of 8 weeks of the treatment duration will be based on the fact that the robust eﬀects of acupuncture in cancer patients will be generally observed within 8 weeks of treatment.

SUMMARY:
Elderly cancer patients would suffer cognitive impairment due to chemotherapy, and a series of neurocognitive symptoms, known as "chemobrain". Chinese acupuncture plus herbal decoctions is an emerging therapeutic option for chemotherapy induced cognitive impairment in elderly cancer patients, despite limited supporting evidence. By evaluating this novel Chinese medicine mode in elderly cancer patients at our institution, the investigators aim to contribute to the existing knowledge in this area while establishing a basis for further research.

The investigators will perform a study of all cases of "chemobrain" related elderly cancer patients treated with Chinese acupuncture from 2023 to 2025. The investigators would enroll 168 elderly cancer patients with clinically confirmed chemobrain; those for Chinese acupuncture will be treated with electroacupuncture (2 sessions per week over 8 weeks) ; the others will be received conventional drug therapy, or palliative-intent therapy. The Montreal Cognitive Assessment (MoCA) will be served as the primary outcome. Digit span test will be the secondary outcome for attentional function and working memory. The quality of life and multiple functional assessments will also be evaluated.

DETAILED DESCRIPTION:
Elderly cancer patients would suffer cognitive impairment due to chemotherapy, and a series of neurocognitive symptoms, known as "chemobrain". Chinese acupuncture plus herbal decoctions is an emerging therapeutic option for chemotherapy-induced cognitive impairment in elderly cancer patients, despite limited supporting evidence. By evaluating this novel Chinese medicine mode in elderly cancer patients at our institution, the investigators would like to contribute to the existing knowledge in this area while establishing a basis for further research.

This randomized controlled trial would be conducted from Jan 2023 to December 2025 in clinics of Nanjing 1st Hospital, Nanjing, China. Potentially eligible patients will be recruited through clinical oncologists' referral from local hospital and advertisement. The study protocol should be approved by Institutional Review Board(IRB) of the Nanjing 1st Hospital. The investigators will enroll 168 elderly cancer patients with clinically confirmed chemobrain.

Acupuncture intervention will be conducted for 2 sessions per week over 8 consecutive weeks. The determination of 8 weeks of the treatment duration will be based on the fact that the robust eﬀects of acupuncture in cancer patients will be generally observed within 8 weeks of treatment.

The primary outcome will be measured using the Montreal Cognitive Assessment(MoCA) which has been extensively used in the study of cognitive disorders. The forward and reverse digit span test would serve the secondary outcomes to detect attentional function and working memory. In addition, EORTCQLQ-C30 will be used to examine the quality of life of elderly cancer patients. Functional changes and side eﬀects associated with therapies will be measured using the Functional Assessment of Cancer Therapy (FACT), Functional Assessment of Chronic Illness Therapy (FACIT), Functional Assessment of Anorexia/Cachexia Therapy (FAACT), Functional Assessment of Cancer Therapy-Taxane (FACT-Taxane), and Functional Assessment of Cancer Therapy-Biologic Response Modiﬁer (FACT-BRM). These instruments have been widely used in elderly cancer patients. Most items of these functional assessments are 5-point Likert scale questions. Functional items which would be rated as "3" (quite a bit) or higher and incidences would be signiﬁcantly diﬀerent between the two groups in any assessment point will be extracted for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly cancer patients >60 years old;
2. Patients clinically confirmed with malignant tumor ;
3. Chemotherapy related cognitive impairment anticipated.

Exclusion Criteria:

1. Chemotherapy received in the past two years;
2. Implanted pacemaker in the body and epilepsy or other unstable diseases.
3. Participated in drug research within the past six years;
4. Alcohol or drug abuse in the past years;
5. Fear of needles;
6. History of stroke or head trauma;
7. Have a history of mood disorders or mental illness.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in score on MoCA | Baseline, Week 2, Week 4, Week 6, Week 8
  The primary outcome will be measured using the Montreal Cognitive Assessment(MoCA)
The incidences of adverse events | up to Week 8
  The incidences of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao S, Zhang J, Wan H, Tao C, Hu M, Liang W, Xu Z, Xu B, Zhang J, Wang G, Li P, Lyu G, Gong Y. Role of Chinese Acupuncture in the Treatment for Chemotherapy-Induced Cognitive Impairment in Older Patients With Cancer: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 8;13:e53853. doi: 10.2196/53853. PMID 38329790